CLINICAL TRIAL: NCT00770575
Title: Double Blinded Study of the Effects of Pioglitazone in Combination With Atorvastatin in Comparison to Atorvastatin Treatment Alone on Intima-Media Thickness in Patients at Risk for Vascular Complications
Brief Title: Efficacy Study of Pioglitazone and Atorvastatin Combination Therapy in Treating Subjects With Elevated Risk for Cardiovascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma GmbH, Aachen (Germany)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATS K015; 2004-004463-30 (EudraCT Number); D-PIO-106 (Other: Takeda ID); U1111-1115-9124 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Cardiovascular Diseases
Keywords: Biological Markers; Biochemical Markers; Carotid Artery, Internal; Carotid Artery, Common; Marker, Surrogate; Vascular Diseases; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases; Diabetes Mellitus | interventions — Pioglitazone; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone 30mg to 45 mg QD + Atorvastatin 20 mg to 40 mg QD (Experimental)
  Interventions: Drug: Pioglitazone and atorvastatin
- Atorvastatin 20mg to 40 mg QD (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pioglitazone and atorvastatin — Pioglitazone 30 mg, capsules, orally, once daily and atorvastatin 20 mg, tablets, orally, once daily for 4 weeks; increase to:
  Pioglitazone 45 mg, capsules, orally, once daily and atorvastatin 40 mg, tablets, orally, once daily for up to 20 weeks.
  Other Names: ACTOS®; AD4833
  Arms: Pioglitazone 30mg to 45 mg QD + Atorvastatin 20 mg to 40 mg QD
Drug: Atorvastatin — Pioglitazone placebo-matching capsules, orally, once daily and atorvastatin 20 mg, tablets, orally, once daily for 4 weeks; increased to
  Pioglitazone placebo-matching capsules, orally, once daily and atorvastatin 40 mg, tablets, orally, once daily for up to 20 weeks.
  Arms: Atorvastatin 20mg to 40 mg QD

SUMMARY:
The purpose of this study is to determine the effect of pioglitazone, once daily (QD), and atorvastatin combination therapy compared to atorvastatin monotherapy in patients at risk for cardiovascular disease.

DETAILED DESCRIPTION:
Carotid intima-media thickness is a well described surrogate marker for cardiovascular risk. A thickened carotid intima media layer correlates not only with the presence of cardiovascular risk factors but also the risk of future macrovascular events such as myocardial infarction and stroke. The interventional approach of cardiovascular risk factors with angiotensin converting enzyme system blockers, calcium antagonists or beta blockers can result in reduction of progression or even net regression of carotid intima-media thickness. The most potent agents, however, are statins which have consistently shown effects on carotid intima-media thickness in patients with hypercholesterolemia and/or atherosclerotic disease.

Peroxisome proliferator activator receptor-gamma activation by thiazolidinediones is a promising new approach which reduces insulin resistance and improves lipid profile. In addition to their metabolic activities, peroxisome proliferator activator receptor-gamma activators were shown to exert anti-inflammatory effects, to improve endothelial function and to inhibit atherogenesis in diabetic and in non-diabetic atherosclerosis-prone animal models. Treatment with peroxisome proliferator activator receptor-gamma agonists have shown to reduce arterial pressure and carotid intima-media thickness in diabetic and non-diabetic patients at risk for cardiovascular disease.

The aim of this study is to evaluate the effect of Pioglitazone in addition to Atorvastatin compared to Atorvastatin alone on vascular risk markers and intima-media thickness in patients with elevated risk for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Intima-media thickness of Common Carotid Artery greater than or equal to 0.8 mm (at least on one side).
* Increased cardiovascular risk defined as one or more of the following:

  * medical history of infarction
  * coronary angiography with proven cardiovascular disease
  * instable Angina pectoris
  * duplex-sonography of cervical or leg vessels with proven atherosclerotic vascular alterations
  * electrocardiogram with ischemia
  * stroke
  * transient ischemic attack
  * peripheral arterial occlusion
  * vessel surgery
  * hypertension (RR greater than 140/90)
  * antihypertensives
  * high density lipoprotein less than 40 mg/dl.
* Body mass index greater than or equal to 25 kg/m2.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* History of overt type-2-diabetes according to the World Health Organization criteria.
* History of type-1-diabetes.
* History of more than one unexplained hypoglycemic episode within the last 6 months.
* Statin therapy within the last 4 weeks.
* Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures.
* History of severe or multiple allergies.
* Treatment with any other investigational drug within 3 months before trial entry.
* Progressive fatal disease.
* Myopathy.
* Drug or alcohol abuse within the last 5 years.
* Smoker defined as patient with evidence or history of tobacco or nicotine use within the last 6 months before the screening visit.
* A history of heart failure (New York Heart Association stage II - IV) or significant respiratory, gastrointestinal, hepatic (glutamate-pyruvate-transaminase time greater than 2.5 times the normal reference range), renal (creatinine greater than 2.0 mg/dl) or hematological disease.
* Blood donation within the last 30 days.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * ciclosporin
  * erythromycin
  * clarithromycin
  * itraconazole
  * ketoconazole
  * nefazodone
  * niacin
  * gemfibrozil and other fibrates
  * HIV-Protease-Inhibitors
* Pre-treatment with thiazolidinediones within 3 months before trial entry.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2005-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change in the intima-media thickness of the common carotid artery. | Week 24.

SECONDARY OUTCOMES:
Change in the intima-media thickness of the internal carotid artery. | Week 24.
Change in the intima-media thickness of the carotid bulbus. | Week 24.
Change from Baseline in Efficacy Laboratory findings (Interleukin-6, high sensitive C reactive peptide and monocyte chemotactic protein-1) | Week: 24.
Change from Baseline in Efficacy Laboratory findings (matrix metalloproteinase-9, soluble CD40 Ligand, P-Selectin, soluble intracellular adhesion molecule 1 and soluble vascular cell adhesion molecule 1). | Week: 24.
Change from Baseline in Efficacy Laboratory findings (adiponectin, tissue plasminogen activator, Plasma glucose, Insulin and Intact proinsulin). | Week: 24.
Change from Baseline in Efficacy Laboratory findings (blood lipids (total cholesterol, high density lipoprotein, triglycerides) and low density lipoprotein-subfractions). | Week: 24.
Change from Baseline in Glycosylated Hemoglobin. | Week: 24.
Change from Baseline in Beta cell function (Homeostatic Model Assessment - beta cell response Score). | Week: 24.
Change from Baseline in Insulin sensitivity using the Homeostatic Model Assessment - Sensitivity Score). | Week: 24.
Change from Baseline in Microcirculation assessment. | Week: 24.
Change from Baseline in Pulse wave velocity. | Weeks: 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Research/Licensing/New Products, Study Director — Takeda Pharma Gmbh, Aachen (Germany)

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI